CLINICAL TRIAL: NCT06826287
Title: More Than Cerebral Cortex: 7T Anatomo-functional Characterization of Cortical, Subcortical, and Cerebellar Structures Involved in THE Network of Action Observation
Brief Title: 7T Anatomo-functional Characterization of Structures in the Action Observation Network
Acronym: 7T-ATHENA
Status: Recruiting | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Collaborators: University of Parma (Other); Fondazione IMAGO7 (Unknown)
Responsible Party: Sponsor
Other Study IDs: 7T-ATHENA
Record Dates: First submitted 2025-01-22; First posted 2025-02-13 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Brain Function; Cerebral Palsy
Keywords: magnetic resonance imaging; ultra high field; action observation network; cerebral palsy; functional re-organization; neural plasticity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy Controls: Subject without any known neurological and psychiatric pathologies
  Interventions: Other: 7T MR exam
- CP patients: Patients with pre-, peri- or post-natal brain injury, as documented in a previous brain MRI examination
  Interventions: Other: 7T MR exam; Other: clinical assessment

INTERVENTIONS:
Other: 7T MR exam — a 7 Tesla MRI scan, with a functional and anatomical dedicated protocol
Other: clinical assessment — A comprehensive clinical assessment before the MRI exam.
  Groups: CP patients

SUMMARY:
The goal of this study is to explore the anatomical-functional characteristics of the AON circuit (with particular interest for subcortical areas and the cerebellum), and the cortico-subcortical connectivity of the nodes of the AON circuit, using an ultra-high field (7T), high spatial resolution Magnetic Resonance Imaging protocol.

The main questions it aims to answer are:

* Can we demonstrate the involvement of subcortical areas and cerebellum in the AON circuit in each single-subject?
* Can we obtain similar results in a small group of patients with Cerebral Palsy (CP), in order to demonstrate the feasibility of this approach for the study of the mechanisms of AON reorganization, after early brain damage?
* Are different patterns of functional activation correlated to different clinical characteristics of CP patients?

Participants will perform a 7 Tesla MRI scan, with a functional and anatomical dedicated protocol and will have a comprehensive clinical assessment before the MRI exam.

DETAILED DESCRIPTION:
In healthy humans, brain functional representation of actions, either executed or observed, relies on the human action observation network (AON). Several studies demonstrated that AON activation is crucial for action understanding and for subserving imitation by observation of new motor skills. The demonstration of the activation of this circuit in patients with motor disorders have opened the way to new rehabilitation protocols based on the observation of meaningful actions followed by their execution (Observation to Imitate), often referred as Action Observation Therapy (AOT). In the last decade, AOT was widely used in adult stroke patients as well as in children with cerebral palsy (CP). Overall, these studies demonstrate a significant motor improvement after therapy, that is maintained at follow-up.

Functional Magnetic Resonance Imaging (fMRI) studies on the effects of AOT found a positive correlation between the functional improvements of manual abilities of these patients and the enlargement of movement-related brain regions, suggesting that AOT can promote the activation of mechanisms of brain plasticity and functional reorganization of the cortical areas responsible for movements. Recently, fMRI studies have demonstrated that also other brain regions, such as the cerebellum, the thalamus and the basal ganglia, belong to the AON.

Despite numerous studies on AON, the fine-grained details of this complex network, especially at subcortical level, and the reciprocal interactions between different brain regions are largely unknown. Moreover, no studies are available at submillimeter level concerning the involvement of subcortical structures. Compared with lower magnetic field systems, Ultra-High Field Magnetic Resonance (UHF-MR) permits a remarkable gain in terms of signal to noise ratio (SNR). This significant increase in SNR produces a great improvement of all imaging parameters, and can be exploited increasing spatial and/or temporal resolution. Moreover, at 7T, we assist also to an empowered sensitivity of the signal to modifications of the composition of tissue that can be translated in new or improved contrasts, such as susceptibility-weighted imaging.

fMRI technique is an advanced MR method that benefits from the use of UHF thanks to the positive combination of increased SNR and increased sensitivity to the effect generating the contrast (BOLD effect).

It has been demonstrated that an increase in the spatial resolution of UHF fMRI allows to describe the functional architecture of the cerebral cortex at mesoscopic (sub-millimeter) scale, hence revealing cortical columns-laminar fMRI profiles, and to segment subcortical structures, to explore their functional selectivity to external stimuli and topographic organization, and to study the cortex. Moreover, the increase in the sensitivity of fMRI at 7T allows to obtain statistically significant functional maps of brain activation not only in groups of subjects but also in individual subjects and individual events, opening new perspectives in the use of fMRI for clinical purposes.

The present study aims to use 7T fMRI to understand the mechanisms of the functional organization of the AON circuit, and in particular the relationship between the cerebral cortex and other structures such as the subcortical nuclei and the cerebellum, and to explore how this organization changes in the presence of lesions acquired at an early age, such as in patients with brain lesions that arose in the pre- or perinatal period, like Cerebral Palsy (CP).

We intend to enroll 28 healthy human subjects and 12 adolescents or young adults with CP. All participants will perform a 7 Tesla MRI scan, with a functional and anatomical dedicated protocol and CP patients will have a comprehensive clinical assessment before the MRI exam.

The MR protocol includes 3D MR sequences with very high spatial resolution. In particular, T1-weighted sequences with isotropic voxel size of 0.8mm is used in order to highlight and segment small substructures, but at the same time evaluating the compliance of subjects, especially of patients, in maintaining the position for long acquisition, without introducing motion artifacts. Analogously, 3D FLAIR sequences are acquired for a detailed study of lesions in CP patients.

fMRI acquisitions in humans are carried out by using Gradient-Echo Echo-Planar Imaging (GRE-EPI) sequences with spatial resolutions depending on the target of each functional series and by using imaging acceleration techniques as SENSE and multi-band approaches. For the study of functional connectivity and the whole AON circuit, comprehensive of the cerebellum, we will privilege whole brain coverage and relatively short temporal resolution (1-1.5 seconds), with a spatial resolution of 1.5mm isotropic voxel. On the other hand, for small substructures and laminar column studies, we will optimize an fMRI acquisition with isotropic voxel size of 0.7-0.9mm.

As functional task we use paradigms already described in previous studies and adapted for the 7T scanner.

Visual stimuli are presented in binocular vision by means of Liquid Cristal Display (LCD) goggles (VisuaStim-SVGA-Resonance Technology, USA). Participants observe short video-clips (lasting 4 s each), showing unimanual or bimanual actions performed by an actor, from a subjective perspective. The observed actions consist in grasping and using different tools (e.g., hammering, using a screwdriver, opening a jar etc.) or, as control condition, observation of the static initial frame of each clip. The objects are of different colors in order to avoid visual adaptation. The visual characteristics of each video are balanced between the experimental conditions to control the effects of brightness, contrast, sharpness and amount of visual information. During the rest period, in the absence of experimental stimuli, the participant have to fixate a white cross on a black background. During the entire fMRI acquisition, subject's performance are visually checked by the experimenter and kinematic parameters are recorded by using MR-compatible cameras.

ELIGIBILITY:
For CP patients

Inclusion Criteria:

* Patients with pre-, peri- or post-natal brain injury, documented by a previous MRI examination of the brain;
* Intellectual development within the norm or within the mild deficit area, to guarantee understanding and cooperation in the 7T fMRI study;
* Understanding of the Italian language;

Exclusion Criteria:

* Contraindications to performing the 7T fMRI exam;
* Neuropsychiatric comorbidity that precludes collaboration in the 7T fMRI study;
* Lack of capacity to understand and to will;
* Pregnancy;

For Healthy Controls

Inclusion Criteria:

* Absence of known neurological and psychiatric pathologies;
* Understanding of the Italian language;

Exclusion Criteria:

* Contraindications to performing the 7T fMRI exam;
* Neuropsychiatric comorbidity that precludes collaboration in the 7T fMRI study;
* Lack of capacity to understand and to will;
* Pregnancy;

Ages: 11 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: primary care clinic for CP; community sample for HC.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2025-08-09 (Estimated); Study Completion 2025-08-09 (Estimated)

PRIMARY OUTCOMES:
7T activation maps of the AON | Day 0
  volume (in cubic millimeters), coordinates (in millimeters), and percentage of signal change of the cortical, subcortical and cerebellar areas elicited by the observation of goal-directed actions
7T connectivity maps of the AON | Day 0
  correlation between each pair of the cortical, subcortical and cerebellar areas elicited by the observation of goal-directed actions

SECONDARY OUTCOMES:
reproducibility | Day 0
  percentage of healthy subjects in which it is possible to identify the AON circuit
clinical correlation | Day 0
  correlation between characteristics of activations (described as primary outcomes) and clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Laura Biagi, PhD, Principal Investigator — IRCCS Stella Maris
Locations (2):
- Italy (2):
  - Fondazione IMAGO7, Calambrone, PISA
  - IRCCS Fondazione Stella Maris, Calambrone, Pisa

IPD SHARING:
Plan to Share IPD: Undecided
To be decided, verifying the compliance with European General Data Protection Regulation (GDPR) law